CLINICAL TRIAL: NCT04088552
Title: Preventing Chronic Disease (HIV, Diabetes, Hypertension, Obesity) Among Older Hispanic Women in Broward
Brief Title: Preventing Chronic Disease: ActuaYa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Community Foundation of Broward (Unknown)
Responsible Party: Principal Investigator, Rosina Cianelli, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20190373
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ActuaYa Arm (Experimental): Participants will receive educational sessions, facilitated discussions and an exercise program.
  Interventions: Other: Go4Life-Physical Activity/Exercise Program "Workout to Go" 5; Behavioral: ActuaYa Educational Sessions

INTERVENTIONS:
Other: Go4Life-Physical Activity/Exercise Program "Workout to Go" 5 — The Go4Life-Physical Activity/Exercise Program "Workout to Go" 5 Program is an exercise regimen provided to participants. Participants will be provided a booklet with exercise routines that requires minimal equipment and can be performed anywhere for approximately 30 minutes per session. Recommendation on staying active by increasing daily steps through walking will also be recommended as part of the regimen.
Behavioral: ActuaYa Educational Sessions — The ActuaYa Educational Sessions will be delivered by a facilitator in 3 separate sessions with each session lasting 2.5 hours for a total of 7.5 hours administered for the study duration. Each session will be conducted in separate groups of 6-10 participants. Session 1 will discuss the impact of chronic disease in the older Hispanic community. Session 2 will discuss the communication and negotiation with the family and partner. Session 3 will discuss saying goodbye and having a plan for a healthy lifestyle.

SUMMARY:
The purpose of the study is to help older Hispanic women to increase physical activity, reach a healthy body weight, increase self-esteem and mood and increase knowledge about chronic diseases such as hypertension, diabetes, and HIV.

ELIGIBILITY:
Inclusion Criteria

1. Must self-identify as a Hispanic woman
2. Must be aged 50 years or older
3. Must not already be engaging in exercise for >150 minutes per week
4. Must be able to ambulate without the use of assistive devices
5. Must have an intelligent phone iOS or Android
6. Must be willing and able to participate in the informed consent process.

Exclusion Criteria

1. Participants that do not meet the above-mentioned criteria.
2. In the opinion of the investigator, have any clinical condition that would make the participant unsuitable to participate.
3. Participants who are currently participating in another investigational study.
4. Participants that need a medical clearance for exercise based on the American College of Sports Medicine exercise participation algorithm.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Change in mean Hemoglobin A1C (HbA1c) levels | Baseline, 6 months
  HbA1c will be measured from finger stick blood sample.
Change in Blood Pressure | Baseline, 6 months
  Changes in blood pressure will be measured using a manual sphygmomanometer by a registered nurse.
Change in Body Mass Index (BMI) | Baseline, 6 months
  BMI will be measured by weight and height using the formula: 703 multiplied by the weight in lbs divided by the square of height in inches.
Change in self-efficacy for condom use | Baseline, 6 months
  Measured using the HIV self-efficacy for condom use survey. Scores range from 7-28. A higher score indicates a higher level of self-efficacy for condom use.
Change in nutritional habits | Baseline, 6 months
  Change in nutritional habits will be evaluated via the Healthy Eating Index (HEI) using the self-reported data from the nutrition survey. The HEI scores range from 0 to 100 with a higher score indicating healthier eating habits with food intake aligning with key dietary recommendations from the Dietary Guidelines for Americans.
Change in active lifestyle as assessed by daily steps | Baseline, 6 months
  Change in active lifestyle will be assessed by the amount of daily steps taken as assessed using a study provided wrist pedometer.
Change in active lifestyle as assessed by a self-report log | Baseline, 6 months
  Change in active lifestyle will be assessed by the number of days per week the participant completed the recommended 30-minutes exercise via a self-report log.
Change in active lifestyle as assessed by the Exercise Survey | Baseline, 6 months
  Change in active lifestyle will be assessed using the Exercise Survey. The exercise survey is a 19-item survey with each item having a score ranging from 0-10. A higher total score indicates a higher level of physical activity.
Change in active lifestyle as assessed by the Exercise Question Survey | Baseline, 6 months
  Change in active lifestyle will be assessed using the Exercise Question Survey. The exercise survey is a 9-item survey with total score ranging from 0-90. A higher total score indicates a higher level of physical activity.
Change in HIV risk behaviors | Baseline, 6 months
  Change in HIV risk behaviors will be assessed using the Partner Table Survey. The Partner Table Survey is a 5-item survey with a total score ranging from 1-17 with a higher score indicating a higher HIV risk behavior.
Change in body fat composition | Baseline, 6 months
  Measured using a bioelectrical impedance analysis.
Change in abdominal circumference | Baseline, 6 months
  Measured using a measuring tape.

SECONDARY OUTCOMES:
Change in knowledge regarding obesity | Baseline, 6 months
  Change in knowledge regarding obesity will be measured using the obesity knowledge and risk perception questionnaire. For obesity knowledge, the scores range from 6-12. A higher score indicates a lower level of obesity-related knowledge.
Change in risk perception regarding obesity | Baseline, 6 months
  Change in risk perception regarding obesity will be measured using the obesity knowledge and risk perception questionnaire. For obesity risk perception, the scores range from 3-9. A higher score indicates a lower level of obesity risk perception.
Change in knowledge regarding diabetes | Baseline, 6 months
  Change in diabetes knowledge will be measured using the Diabetes Knowledge Questionnaire (DKQ-24). It is a 24 item questionnaire wherein a score of 17 or more correct responses indicate sufficient diabetes knowledge and a score of 6 or less correct responses indicate insufficient diabetes knowledge.
Change in HIV knowledge | Baseline, 6 months
  Change in HIV knowledge will be measured via the HIV Knowledge Scale. The score ranges from 0-12 with a higher score indicating a higher level of HIV-related knowledge.
Change in HIV risk perception | Baseline, 6 months
  Change in HIV risk perception will be measured via the HIV Risk Perception Scale. The total score ranges from 4-14 with a higher score indicating a higher level of HIV-related knowledge.
Change in self-esteem | Baseline, 6 months
  Change in self-esteem will be measured by the Rosenberg Self-Esteem Scale via interview. The total score ranges from 0 to 30 with a score of 14 and less indicating low self-esteem.
Change in depressive symptoms as assessed by the CES-D20 | Baseline, 6 months
  Change in depressive symptoms will be measured using the Center for Epidemiologic Studies Depression Scale (CES-D20). The CES-D20 has a total score ranging from 0 to 60 with a higher score indicating greater depressive symptoms.
Change in depressive symptoms as assessed by the GDS | Baseline, 6 months
  Change in depressive symptoms will be measured using the Geriatric Depression Scale (GDS). The GDS has a total score ranging from 0-15 with a higher score indicating higher depressive symptoms. A score of 6 to 9 indicates suggestive depressive symptoms and a score of 10 to 15 indicates depressive symptoms.
Change in health care related habits | Baseline, 6 months
  Change in healthcare related habits is measured via the Health Care-Related Factors Questionnaire. The total score ranges from 26 to 43 with a higher score indicating lesser health care related habits.
Change in technology use | Baseline, 6 months
  Change in technology use will be measured using a questionnaire assessing ability to use technology (pedometer, smartphones, apps, internet). The total score ranges from 13-26 with a higher score indicating a lower ability to use technology.
Change in knowledge regarding hypertension | Baseline, 6 months
  Change in knowledge regarding hypertension is measured using the Hypertension Survey. The Hypertension Survey is a 10-item survey with a totals score ranging from 0-10 with a higher score indicating increased knowledge regarding hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Rosina Cianelli, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No